CLINICAL TRIAL: NCT06718231
Title: Transcutaneous Electrical Acupoint Stimulation Alleviate Postoperative Depression in Video-assisted Thoracoscopic Surgery: a Randomized Controlled Trial
Brief Title: TAES Alleviate Post-VATS Depression
Acronym: TAES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fuling Central Hospital of Chongqing City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TAES for VATS depression
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Depression After Video-assisted Thoracoscopic Surgery
Keywords: Transcutaneous electrical acupoint stimulation (TAES); depression; video-assisted thoracoscopic surgery; interleukin-6; tumor necrosis factor-α
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The traditional Chinese medicine doctor will administer the intervention based on the randomized grouping to ensure the double-blind nature of the study. Neither anesthesiologists nor outcome assessors will aware of patient randomization. The participants will be blinded with reference to Song et al.'s study. In TAES group, electrode pads will be fixed on the bilateral HT7 (Shenmen), PC6 (Neiguan), LI4 (Hegu), LU5 (Chize) and Extra (Anmian), the current set based on the participants ' maximum tolerance and muscle fibrillation. In the Sham-TAES group, electrodes will be fixed at 4 cm interior to the bilateral Shenmen, Neiguan, Hegu, Chize, and Anmian acupoints , and the frequency current setting given in the same way as in the TAES group to make the patients think that they received the TAES treatment. Therefore, all participants will be unaware of randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Active Comparator): the electrodes will be fixed at acupointsShenmen,Neiguan,Hegu,Chize,Anmian bilaterally
  Interventions: Behavioral: Transcutaneous electrical acupoint stimulation
- Group S (Sham Comparator): the electrode pads will be fixed at the bilateral sham acupoints
  Interventions: Behavioral: Sham-TAES

INTERVENTIONS:
Behavioral: Transcutaneous electrical acupoint stimulation — After entering the operating room, an experienced traditional Chinese medicine doctor will locate the bilateral Shenmen, Neiguan, Hegu, Chize, and Anmian acupoints, and sham acupoints. The target treatment acupoints will be wiped with 75% ethanol, and after the ethanol had evaporated, electrode pads (50 × 50 mm) will be placed and fixed according to the different groups. Thirty minutes before anesthesia, a TAES stimulator (Hwato Electronic Acupuncture Treatment Instrument, model no: SDZ-III; Suzhou Medical Appliances Co. Ltd, Suzhou, China) will be connected with a frequency setting of 2/10 Hz (2 Hz for 10 s and 10 Hz for 5 s), in dense-disperse mode. The current intensity will be set according to the patient's maximum tolerance and muscle twitching and continued until the end of the surgery.
  Arms: Group T
Behavioral: Sham-TAES — After entering the operating room, an experienced traditional Chinese medicine doctor will locate the bilateral sham acupoints. The Sham acupoints is 4 cm interior to the bilateral Shenmen, Neiguan, Hegu, Chize, and Anmian acupoints. The sham acupoints will be wiped with 75% ethanol, and after the ethanol had evaporated, electrode pads (50 × 50 mm) will be placed and fixed according to the different groups. Thirty minutes before anesthesia, a TAES stimulator (Hwato Electronic Acupuncture Treatment Instrument, model no: SDZ-III; Suzhou Medical Appliances Co. Ltd, Suzhou, China) will be connected with a frequency setting of 2/10 Hz (2 Hz for 10 s and 10 Hz for 5 s), in dense-disperse mode. The current intensity will be set according to the patient's maximum tolerance and muscle twitching and continued until the end of the surgery
  Arms: Group S

SUMMARY:
Depression can significantly affect postoperative rehabilitation quality and increase the mortality of patients who receive video-assisted thoracoscopic surgery (VATS). This study intend to evaluate the transcutaneous electrical acupoint stimulation (TEAS) of VATS safety and the efficacy of the postoperative depression compared to a sham group.

DETAILED DESCRIPTION:
Depression is a common psychiatric problem in perioperative period in patients who receive video-assisted thoracoscopic surgery (VATS). Multiple research have pointed out that the incidence of postoperative depression can be as high as 11.8%-34% . Brian et al.reported that the iIncidence of new depressive episodes one year after VATS was as high as 12.4%. Depression not only reduces treatment compliance and quality of life, prolongs hospital stays, and increases postoperati''ve mortality, but can also exacerbate pain and reduce sleep quality, significantly affecting postoperative recovery .

Modern studies report that surgical trauma, pain, sleep disorders, and stress responses increases inflammatory factors such as TNF-α and IL-6, and cause inflammation. This results in a decrease in the production of the monoamine neurotransmitters serotonin and norepinephrine in the brain, which causes depression. Therefore, the antidepressant drugs widely used in clinical practice are serotonin reuptake inhibitors; however, they are not only expensive and slow to act, but also have various side reactions, such as decreased libido, sexual dysfunction, headache, gastrointestinal symptoms, irritability, and anxiety. Further, long-term use may also cause damage to the nervous system.

Transcutaneous acupoint electrical stimulation (TAES) is an innovative diagnostic and therapeutic technique used in traditional Chinese medicine that integrates transcutaneous nerve electrical stimulation with meridian acupoints. It offers numerous advantages, such as being noninvasive, painless, simple to operate, with high treatment compliance, and minimal side effects. Multiple studies have shown that TAES not only has analgesic, anti-stress, and anti-inflammatory effects and can improve postoperative sleep disorders but can also directly increase the concentration of serotonin in the brain. Therefore, TAES may effectively improve post-VATS depression symptoms. This prospective, randomized, controlled, double blind, single-arm, single-center study will provide insights oninto the safety and effectiveness of TAES in improving post-VATS.

ELIGIBILITY:
Inclusion Criteria:

Unilateral VATS performed under general anesthesia due to pulmonary nodules; The age ranged from 18 to 65 years; American Society of Anesthesiologists (ASA) classification II-III; The patient has normal consciousness, with no facial paralysis, is capable of cooperating with treatment, and provides signed informed consent.

Exclusion Criteria:

Merge the skin of local acupoint infectors; Patients with upper extremity nerve injury; Patients with implanted pacemakers; Alcoholism or long-term use of opioid, hormonal, and anti-inflammatory analgesics; Allergic to the drug used in the study; Those who recently received TAES or acupoint treatment; Patients with history of psychiatric disorders or current use of psychiatric medication; Receiving treatment with monoamine oxidase inhibitors; Severe disease of the heart, brain, liver, kidneys, or hematopoietic system; Patients unable to cooperate with the study for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory score 30 days postoperatively | 30 days postoperatively
  The self-rating Scale for Depression consists of 21 groups of questions, each group has 4 statements, and each sentence corresponds to an Arabic numeral.Participants choose the statement that best suits their situation according to their own feeling.After all 21 groups have been completed, the total score of each group is added

SECONDARY OUTCOMES:
Beck Depression Inventory score 2 days postoperatively | 2 days postoperatively
  The self-rating Scale for Depression consists of 21 groups of questions, each group has 4 statements, and each sentence corresponds to an Arabic numeral.Participants choose the statement that best suits their situation according to their own feeling.After all 21 groups have been completed, the total score of each group is added
Serum Interleukin-6 concentration 2 days after surgery | 2 days after surgery
  Enzyme-linked immunosorbent assay was used to measure serum interleukin-6 concentration 2 days after surgery
Serum tumor necrosis factor-α concentration 2 days after surgery | 2 days after surgery
  Enzyme-linked immunosorbent assay was used to measure serum tumor necrosis factor-α concentration 2 days after surgery
24h postoperative resting pain numerical rating scale (NRS) score | 24 hours after surgery
  The Numeric Rating Scale is used to assess pain.Ask participant to rate based on how they feel pain.0 is painless and 10 is the most severe pain
48h postoperative resting pain numerical rating scale (NRS) score | 48 hours after surgery
  The Numeric Rating Scale is used to assess pain.Ask participant to rate based on how they feel pain.0 is painless and 10 is the most severe pain
24h postoperative moving NRS pain score | 24 hours after surgery
  The Numeric Rating Scale is used to assess pain.Ask participant to rate based on how they feel pain.0 is painless and 10 is the most severe pain
48h postoperative moving NRS pain score | 48 hours after surgery
  The Numeric Rating Scale is used to assess pain.Ask participant to rate based on how they feel pain.0 is painless and 10 is the most severe pain
Dosage of patient controlled intravenous analgesia 24h after surgery | 24 hours after surgery
  patient controlled intravenous analgesia record
Dosage of patient controlled intravenous analgesia 48h after surgery | 48 hours after surgery
  patient controlled intravenous analgesia record
Sleep NRS score 2 days after surgery | 2 days after sergury
  A Numeric Rating Scale was used to assess sleep quality. Participants were asked to rate how well they slept. 0 is good sleep and 10 is unable to sleep at all
TAES-related complications | 2 days after sergury
  dermatitis, allergic reactions, dizziness,drowsiness

CONTACTS AND LOCATIONS:
Locations (1):
- Fuling Central Hospital of Chongqing, Fuling, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
To protect patient privacy, we consider keeping the data private.After the study concludes, the raw data and research findings will be reported to the Research Management Committee.the original data will be available from the researchers via email through official channels.

REFERENCES:
- [Result] He Y, Yuan M, He C, Zhu D, Wang F. The Effects of Transcutaneous Acupoint Electrical Stimulation on Cancer-related Fatigue and Negative Emotions in Cancer Patients: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Contrast Media Mol Imaging. 2022 Jul 31;2022:1225253. doi: 10.1155/2022/1225253. eCollection 2022. PMID 35965622
- [Result] Tsay SL, Cho YC, Chen ML. Acupressure and Transcutaneous Electrical Acupoint Stimulation in improving fatigue, sleep quality and depression in hemodialysis patients. Am J Chin Med. 2004;32(3):407-16. doi: 10.1142/S0192415X04002065. PMID 15344424
- [Result] Wang H, Yang BZ, Guo Q, Jing ZY. [Effect of transcutaneous electrical acupoint stimulation combined with epidural labor analgesia on postpartum depression]. Zhen Ci Yan Jiu. 2021 Mar 25;46(3):231-4. doi: 10.13702/j.1000-0607.200249. Chinese. PMID 33798297
- [Result] Chen WY, Li L, Wang HY, Jiang N. [Effects of Transcutaneous Electrical Acupoint Stimulation for Depression in Late Pregnancy and Impacts on Inflammatory Cytokines]. Zhen Ci Yan Jiu. 2018 Jan 25;43(1):44-8. doi: 10.13702/j.1000-0607.160781. Chinese. PMID 29383894
- [Result] Agrawal S, Szmit M, Welna M, Rudnicki J, Agrawal A, Gozdzik W. Transcutaneous electrical acupoint stimulation to reduce opioid consumption in patients undergoing inguinal hernia repair: protocol for a randomized controlled trial. Trials. 2022 Dec 29;23(1):1064. doi: 10.1186/s13063-022-07019-9. PMID 36581999
- [Result] Chen J, Zhang Y, Li X, Wan Y, Ji X, Wang W, Kang X, Yan W, Fan Z. Efficacy of transcutaneous electrical acupoint stimulation combined with general anesthesia for sedation and postoperative analgesia in minimally invasive lung cancer surgery: A randomized, double-blind, placebo-controlled trial. Thorac Cancer. 2020 Apr;11(4):928-934. doi: 10.1111/1759-7714.13343. Epub 2020 Feb 16. PMID 32062864
- [Result] Song B, Chang Y, Li Y, Zhu J. Effects of Transcutaneous Electrical Acupoint Stimulation on the Postoperative Sleep Quality and Pain of Patients After Video-Assisted Thoracoscopic Surgery: A Prospective, Randomized Controlled Trial. Nat Sci Sleep. 2020 Oct 27;12:809-819. doi: 10.2147/NSS.S270739. eCollection 2020. PMID 33154688
- [Result] Ulett GA, Han S, Han JS. Electroacupuncture: mechanisms and clinical application. Biol Psychiatry. 1998 Jul 15;44(2):129-38. doi: 10.1016/s0006-3223(97)00394-6. PMID 9646895
- [Result] Duan D, Tu Y, Yang X, Liu P. Electroacupuncture Restores 5-HT System Deficit in Chronic Mild Stress-Induced Depressed Rats. Evid Based Complement Alternat Med. 2016;2016:7950635. doi: 10.1155/2016/7950635. Epub 2016 Nov 23. PMID 27994633
- [Result] Yan LP, Liu YG, Wu XT, Li SD, Ma C. [Effect of electroacupuncture intervention on N-methyl-D-aspartic acid receptor expression in spinal cord in rats with chronic constrictive injury of the sciatic nerve]. Zhen Ci Yan Jiu. 2013 Oct;38(5):380-5. Chinese. PMID 24308185
- [Result] Qiao LN, Yang YS, Wang JY, Gao YH, Han YJ, Chen SP, Ji CF, Liu JL. [Effects of electroacupuncture at "Futu" (LI 18), etc. on expression of spinal 5-HT 1 AR mRNA, 5-HT 2 AR mRNA and protein in rats with neck incision pain]. Zhen Ci Yan Jiu. 2011 Dec;36(6):391-6. Chinese. PMID 22379782
- [Result] Wu ZJ, Cai RL, He L, Ma Y, Hu WB, Wang KM. [Effects of electroacupuncture stimulation of "Neiguan" (PC 6) and "Shenmen" (HT7) on contents of 5-hydroxytryptamine in hypothalamic paraventricular nucleus region and serum in hyperlipidemia rats with acute myocardial infarction]. Zhen Ci Yan Jiu. 2013 Dec;38(6):482-7. Chinese. PMID 24579363
- [Result] Liu X, Li S, Wang B, An L, Ren X, Wu H. Intraoperative and postoperative anaesthetic and analgesic effect of multipoint transcutaneous electrical acupuncture stimulation combined with sufentanil anaesthesia in patients undergoing supratentorial craniotomy. Acupunct Med. 2015 Aug;33(4):270-6. doi: 10.1136/acupmed-2014-010749. Epub 2015 Apr 29. PMID 25926298
- [Result] Marwaha S, Palmer E, Suppes T, Cons E, Young AH, Upthegrove R. Novel and emerging treatments for major depression. Lancet. 2023 Jan 14;401(10371):141-153. doi: 10.1016/S0140-6736(22)02080-3. Epub 2022 Dec 16. PMID 36535295
- [Result] Ting EY, Yang AC, Tsai SJ. Role of Interleukin-6 in Depressive Disorder. Int J Mol Sci. 2020 Mar 22;21(6):2194. doi: 10.3390/ijms21062194. PMID 32235786
- [Result] Colucci-D'Amato L, Speranza L, Volpicelli F. Neurotrophic Factor BDNF, Physiological Functions and Therapeutic Potential in Depression, Neurodegeneration and Brain Cancer. Int J Mol Sci. 2020 Oct 21;21(20):7777. doi: 10.3390/ijms21207777. PMID 33096634
- [Result] Wei W, Huang X, Zhu J. Effect of Acupoint Therapies on Postoperative Sleep Quality: A Narrative Review. Med Sci Monit. 2023 Feb 10;29:e938920. doi: 10.12659/MSM.938920. PMID 36760099
- [Result] Schinz K, Steigerwald L, Mantsopoulos K, Gostian AO, Traxdorf M, Sievert M, Rupp R, Iro H, Mueller SK. Depression and female gender associated with higher postoperative pain scores after sinonasal surgery. Acta Otolaryngol. 2022 Jan;142(1):73-77. doi: 10.1080/00016489.2021.2012254. Epub 2021 Dec 23. PMID 34939889
- [Result] Sullivan DR, Forsberg CW, Ganzini L, Au DH, Gould MK, Provenzale D, Slatore CG. Longitudinal Changes in Depression Symptoms and Survival Among Patients With Lung Cancer: A National Cohort Assessment. J Clin Oncol. 2016 Nov 20;34(33):3984-3991. doi: 10.1200/JCO.2016.66.8459. Epub 2016 Oct 31. PMID 27996350
- [Result] O'Gara B, Espinosa Leon JP, Robinson K, Schaefer M, Talmor D, Fischer M. New onset postoperative depression after major surgery: an analysis from a national claims database. BJA Open. 2023 Sep 21;8:100223. doi: 10.1016/j.bjao.2023.100223. eCollection 2023 Dec. PMID 37766788
- [Result] Cheng X, Wang H, Diao M, Jiao H. Effect of S-ketamine on Postoperative Quality of Recovery in Patients Undergoing Video-Assisted Thoracic Surgery. J Cardiothorac Vasc Anesth. 2022 Aug;36(8 Pt B):3049-3056. doi: 10.1053/j.jvca.2022.04.028. Epub 2022 Apr 26. PMID 35613989
- [Result] Zhou Jian SX, Xiaoyi H, Xiang L, He L, Junli C. Effects of mecobalamin combined with ropivacaine for intercostal nerve block on the postoperative depression in patients undergoing thoracoscopic surgery. J Xuzhou Med Univ. 2021;41:189-93
- [Result] Gan SL, Long YQ, Wang QY, Feng CD, Lai CX, Liu CT, Ding YY, Liu H, Peng K, Ji FH. Effect of esketamine on postoperative depressive symptoms in patients undergoing thoracoscopic lung cancer surgery: A randomized controlled trial. Front Psychiatry. 2023 Mar 15;14:1128406. doi: 10.3389/fpsyt.2023.1128406. eCollection 2023. PMID 37009103